CLINICAL TRIAL: NCT04266613
Title: Molecular Biomarkers in Renal Transplant Recipients at Higher Risk of Acute Rejection
Brief Title: TruGraf® Testing in High-Risk Kidney Transplant Recipients
Status: Terminated | Type: Observational
Why Stopped: Sponsor Decision
Sponsor: Transplant Genomics, Inc. (Industry)
Collaborators: The Methodist Hospital Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: TGRP03-US003
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-08

CONDITIONS: Kidney Transplant Rejection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Subjects Enrolled: High immune risk transplant recipients who are undergoing routine management under current standard of care
  Interventions: Diagnostic Test: TruGraf® Testing

INTERVENTIONS:
Diagnostic Test: TruGraf® Testing — 5 mL collection PAXgene blood sample
  Other Names: Peripheral blood gene expression profiling

SUMMARY:
This is an observational study to evaluate TruGraf® testing in high immune risk kidney transplant recipients. TruGraf is the first and only non-invasive test approved by Medicare to rule out silent rejection in stable kidney transplant recipients.

ELIGIBILITY:
Inclusion Criteria:

* High immune risk kidney transplant recipients defined by one of the following criteria: either a positive pretransplant donor specific anti-human leukocyte antigen (HLA) antibody, or a pre-transplant panel reactive antibody >75%.
* Recipient of a primary or subsequent deceased-donor or living donor kidney transplantation.
* Stable serum creatinine (current serum creatinine <2.3 mg/dl, <20% increase compared to the average of the previous 3 serum creatinine levels).
* Kidney transplant patients who are at least 30 days post-transplant.

Exclusion Criteria:

* Need for combined organ transplantation with an extra-renal organ and/or islet cell transplant.
* Recipients who do not meet criteria of high-immune risk.
* Recipients of previous non-renal solid organ and/or islet cell transplantation.
* Infection with HIV.
* Infection with BK.
* Patients that have nephrotic proteinuria (urine protein >3 gm/day).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney transplant recipients with high immune risk who are undergoing routine management
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2021-06-23 (Actual); Study Completion 2021-06-23 (Actual)

PRIMARY OUTCOMES:
Clinical Utility of TruGraf Results | 1 year
  Percent of total number of TruGraf results that the PI identified as having clinical utility
Correlation of TruGraf Results | 1 year
  Percent of total number of TruGraf results that the PI identified as being correlated to other clinical results obtained through the standard of care

CONTACTS AND LOCATIONS:
Overall Officials: John Holman, MD, Study Director — Transplant Genomics, Inc.
Locations (1):
- Houston Methodist Research Institute, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marsh CL, Kurian SM, Rice JC, Whisenant TC, David J, Rose S, Schieve C, Lee D, Case J, Barrick B, Peddi VR, Mannon RB, Knight R, Maluf D, Mandelbrot D, Patel A, Friedewald JJ, Abecassis MM, First MR. Application of TruGraf v1: A Novel Molecular Biomarker for Managing Kidney Transplant Recipients With Stable Renal Function. Transplant Proc. 2019 Apr;51(3):722-728. doi: 10.1016/j.transproceed.2019.01.054. Epub 2019 Jan 26. PMID 30979456
- [Background] First MR, Peddi VR, Mannon R, Knight R, Marsh CL, Kurian SM, Rice JC, Maluf D, Mandelbrot D, Patel A, David J, Schieve C, Lee D, Lewis P, Friedewald JJ, Abecassis MM, Rose S. Investigator Assessment of the Utility of the TruGraf Molecular Diagnostic Test in Clinical Practice. Transplant Proc. 2019 Apr;51(3):729-733. doi: 10.1016/j.transproceed.2018.10.024. Epub 2018 Dec 11. PMID 30979457